CLINICAL TRIAL: NCT06172881
Title: Novel Multifocal Soft Contact Lens Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Myoptechs (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, PI, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023W0119
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Distance Visual Acuity (Experimental): Visual acuity will be measured while participant's wear study lenses.
  Interventions: Device: Investigational Contact Lens

INTERVENTIONS:
Device: Investigational Contact Lens — A soft contact lens that will be worn only at the study visit.

SUMMARY:
A single site, open label protocol will be used to evaluate the safety and quality of vision of a novel soft contact lens. Habitual contact lens wearers will be asked to come to the study site for one visit. Ocular health assessments and visual acuity will be completed with both the study lens and without.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Any gender
3. Any racial or ethnic origin
4. 18 - 40 years of age
5. Distance visual acuity with best corrected visual acuity of 20/25 with each eye
6. Habitual soft contact lens wearer with myopia
7. Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the investigator).

Exclusion Criteria:

1. Current or active ocular inflammation or infection as determined by the Investigator.
2. Astigmatism > 0.75 D in either eye
3. History of previous eye surgery
4. Demonstration or history of corneal ectasia or keratoconus.
5. Pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD, MS, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Distance Visual Acuity
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Distance Visual Acuity
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 29.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity
Description: LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision.
Time Frame: 1 day (This is a single visit study)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Distance Visual Acuity
Number analyzed (Participants) | 10
logMAR
  High Contrast Distance Visual Acuity OD | -0.13 (0.08)
  High Contrast Distance Visual Acuity OS | -0.12 (0.09)

ADVERSE EVENTS:
Time Frame: During study visit (about 1 hour)
Arm/Group | Distance Visual Acuity
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT06172881/Prot_SAP_000.pdf